CLINICAL TRIAL: NCT03570411
Title: Evaluating the Clinical Utility of the T-SPOT.CMV Assay for the Prediction of CMV Reactivation Among Pediatric Patients Undergoing Hematopoietic Cell Transplant
Status: Terminated | Type: Observational
Why Stopped: The company that was contracted to conduct study specific testing was sold and new management chose to pursue interests other than CMV.
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Oxford Immunotec (Industry)
Responsible Party: Sponsor
Other Study IDs: SPOTCMV; NCI-2018-01349 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2018-05-31; First posted 2018-06-27 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: CMV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCT Recipient: All participants who meet eligibility criteria and consent to enrollment on study.
  Blood specimens will be collected for the T-SPOT.CMV blood test from HCT recipients over the course of 6 months, starting weekly at Day +1, biweekly starting at Day +45, and monthly starting at day +120.
  The amount of blood collected at each visit will be based on age.
  Interventions: Diagnostic Test: T-SPOT®.CMV Test
- HCT Donor: Approved allogeneic HCT donor for a HCT recipient enrolled on the SPOTCMV protocol
  A blood sample for the T-SPOT.CMV blood test will be collected from the HCT donor prior to transplant
  Interventions: Diagnostic Test: T-SPOT®.CMV Test

INTERVENTIONS:
Diagnostic Test: T-SPOT®.CMV Test — The T-SPOT.CMV test (Oxford Diagnostic Laboratories) measures the strength of T cell responses to CMV specific antigens. Using whole blood samples obtained through a standard blood collection tube, white blood cells (WBC's) are separated and purified. The cells are quantified and placed into specially designed plates where they are challenged with antigens specific to the disease under study. Disease-specific cells responding to these antigens will release immune messenger molecules, called cytokines. We then use chemistry to allow us to visualize those WBCs releasing cytokines (and hence those which react to the antigen), resulting in a spot on the bottom of the plate, corresponding to the footprint of an individual reacting WBC. Finally, we use an automated image analysis system to identify and count each of these spots to give a quantitative readout. That quantitative readout gives us the frequency of responsive disease-specific cells (Oxford Immunotec, 2017).

SUMMARY:
The ability to distinguish allogeneic hematopoietic cell transplantation (allo-HCT) recipients at risk for cytomegalovirus (CMV) reactivation from those who are not is central for optimal CMV management strategies. Measuring this cell mediated immunity has been proposed as a potent tool to predict those patients at highest risk of CMV reactivation and disease. This study will evaluate the ability of the T-SPOT.CMV test to predict Cytomegalovirus (CMV) reactivation in allogeneic hematopoietic cell transplantation (allo-HCT) pediatric recipients.

Primary Objectives:

To evaluate feasibility of T-SPOT.CMV spot count test in allo-HCT pediatric recipients.

To evaluate association of T-SPOT.CMV spot count in the first sample collected after patient has engrafted with subsequent CMV reactivation in allo-HCT pediatric recipients.

Secondary Objectives:

To evaluate the correlation between T-SPOT.CMV spot count in donors with subsequent recipient CMV spot count.

To explore the relationship between recipient T-SPOT.CMV spot counts and subsequent CMV infection related morbidity and treatment outcomes among pediatric all-HCT recipients.

DETAILED DESCRIPTION:
T-SPOT response will be measured using the results from the T-SPOT.CMV blood test in both HCT recipients and HCT donors.

A blood sample for the T-SPOT.CMV blood test will be collected from the HCT donor prior to transplant.

Blood specimens will be collected for the T-SPOT.CMV blood test from HCT recipients over the course of 6 months, starting weekly at Day +1, biweekly starting at Day +45, and monthly starting at day +120.

HCT recipient participant demographic and clinical characteristics will be collected at enrollment. Additional clinical information will be abstracted from the HCT recipient participants medical record during the study follow-up period. This will include information related to transplant history and outcome, infections, antimicrobial exposure, chemotherapy, and laboratory values related to infectious diseases and immunosuppression.

The feasibility of the T-SPOT.CMV spot count test will be evaluated once the first 30 participants enrolled on study reach day +90. If 75% of patients have at least 1 evaluable samples after engraftment (> 75,000 per microtiter wells), we will proceed with enrollment. If more >25% of patients have all their samples deemed not evaluable due to insufficient mononuclear cell count (<75,000 per microtiter wells) the study will be stopped and concluded as not feasible.

ELIGIBILITY:
HCT Recipient Inclusion Criteria

* Less than 18 years old at the time of study enrollment
* Scheduled to receive allogeneic HCT at St Jude Children's Research Hospital
* HCT recipient has a documented seropositive CMV result prior to enrollment OR The HCT recipient is seronegative, but the HCT donor has a seropositive CMV result as documented in the recipient's medical record.

HCT Recipient Exclusion Criteria

* Any condition or therapy that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the study, or impact the outcome of the study.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

HCT Donor Inclusion Criteria

• Approved allogeneic HCT donor for a HCT recipient enrolled on the SPOTCMV protocol

HCT Donor Exclusion Criteria

• Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 94 HCT recipients and 94 HCT Donors of HCT Recipients on study
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
Percentage of the first 30 participants with at least one evaluable sample | Day +90 after transplant
  Percentage of the first 30 participants enrolled on study reach day +90 with at least one evaluable sample will be reported.
Odds ratio of subsequent reactivation | Up to 180 days after enrollment.
  We define the primary endpoint to the T-SPOT CMV count in the first sample collected after patient has engrafted, which is the time point when one establishes his/her post-transplant immunity. If the count in this sample is less than or equal to 100, the participant will be noted as "low response", while an individual with a spot count greater than 100 will be noted as "high response". Odds ratio of having subsequent CMV reactivation between "low response" and "high response" groups will be estimated.

SECONDARY OUTCOMES:
Correlation coefficient of T-SPOT.CMV spot count in donors with subsequent recipient CMV spot count | Up to 180 days after enrollment.
  The correlation coefficient between T-SPOT.CMV spot count in donors (one-time measure) and maximal recipient's CMV spot count will be calculated with Pearson's or Spearman's correlation coefficient.
Odds ratio of morbidity | Up to 180 days after enrollment.
  The odds ratio with 95% CI of morbidity will be reported from multiple logistic regression.
Odds ratio of treatment outcomes | Up to 180 days after enrollment.
  The odds ratio with 95% CI of treatment outcomes will be reported from multiple logistic regression.
Hazard ratio of morbidity | Up to 180 days after enrollment.
  The hazard ratio with 95% CI of morbidity will be reported from Cox regression model.
Hazard ratio of treatment outcomes | Up to 180 days after enrollment.
  The hazard ratio with 95% CI of treatment outcomes will be reported from Cox regression model.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Hijano, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols